CLINICAL TRIAL: NCT01207258
Title: A Randomized Control Trial of Brief Intervention for Problem Drinking and Partner Violence
Brief Title: Brief Intervention for Problem Drinking and Partner Violence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01AA018705-01A1 (NIH)
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Domestic Violence; Alcohol Abuse
Keywords: Motivational Interviewing; Brief Intervention; Intimate Partner Violence; Domestic Violence; Alcohol Abuse
MeSH Terms: conditions — Alcoholism | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Brief Intervention Group (Experimental): Participants randomly assigned to this group receive a brief motivational enhancement therapy intervention group and are assessed at baseline, weekly for 12 weeks, and at 3, 6 and 12 months.
  Interventions: Behavioral: Motivational Enhancement Therapy
- Assessed Control Group (No Intervention): This group does not receive the intervention and is assessed at baseline, weekly for 12 weeks, and at 3, 6 and 12 months.
- No Contact Control Group (No Intervention): This group does not receive the intervention and is assessed only at 3 months.

INTERVENTIONS:
Behavioral: Motivational Enhancement Therapy — 20 minute manual-driven, optionally audio-recorded Motivational Enhancement Training intervention by a MI-trained therapist during their ED visit and a 10-15 minute phone booster at 7 to 10 days.
  Arms: Brief Intervention Group

SUMMARY:
This study is a randomized controlled trial of a brief intervention for women Emergency Department patients with involvement in both Intimate Partner Violence (IPV) and problem drinking (defined as the full spectrum of hazardous, harmful, or dependent drinking). The study is designed to explore the effectiveness of a low-intensity, gender-sensitive brief motivational intervention, delivered by social workers in the Emergency Department setting, in decreasing IPV and episodes of heavy drinking and increasing rates of follow-up with resources. Social work graduate students and/or staff will be trained to provide brief motivational enhancement therapy (MET) intervention for decreasing heavy drinking and IPV-related injury in women Emergency Department patients.

DETAILED DESCRIPTION:
The investigators will enroll a total of 600 eligible consenting women patients who will be randomized to a Brief Intervention Group (BIG) n=240, an Assessed Care Group (ACG) n=240 or to a No Contact Control Group (NCCG) n=120, that is screened for eligibility and provides basic demographic information but has no further contact with researchers until they are assessed for outcomes only at 3 months. All participants will complete an initial Social Health Survey, a form distributed routinely to all patients in the ED which gives patients an opportunity to self-disclose a variety of social and behavioral risks as part of routine care. As part of the study, patients who disclose any IPV or drinking risk will be asked to complete a further screening (CTS2S and AUDIT) to confirm eligibility prior to randomization. The experimental group (BIG) will receive a 20 minute manual driven, optionally audio-recorded MET intervention by a Motivational Interview (MI)-trained therapist during their ED visit and a 10-15 minute phone booster at 7 to 10 days. The BIG and ACG will be assessed at baseline using the Women's Health Interview to identify potential moderators of the intervention and followed weekly for IPV and drinking outcomes using an Interactive Voice Response System (IVRS) for 12 weeks and phone assessments at 3, 6, and 12 months.

Primary outcomes, assessed for all groups at 3 months, will be the number of heavy drinking days and the incidents of IPV in the last month. Secondary outcomes include number of severe IPV incidents and average weekly alcohol consumption. The investigators will also assess likely mediators of the intervention. Protocol for follow-up contact will be determined by a plan developed by the participant and the MET interventionist. Should a participant decide that it is unsafe to be contacted via telephone, she will be given the option to complete any or all follow-up in the ED. Each time the patient is contacted for follow-up, the researcher will ask if the plan for contact has changed and will implement the necessary changes during the subsequent contacts. In addition, participants will be told that they can contact the PI using the contact information provided on the study's consent materials if the plan changes between contacts. Participants will also be asked at each follow-up contact if they are still interested in participating in the Women's Health Study to ensure ongoing consent. They may decide not to continue participation, and do not need to provide a reason for withdrawal from the study.

ELIGIBILITY:
Inclusion Criteria:

* Registered as an ED patient.
* Able to participate verbally in an English language interview.
* Able to participate cognitively in an English language interview.
* Heavy drinking as assessed by the AUDIT.
* Positive screen for Intimate Partner Violence in the past 3 months.

Exclusion Criteria:

* Intoxication at the time of screening.
* Cognitive impairment or psychosis identified on physical exam or chart review.
* Serious current medical illness or injury, defined as respiratory distress, hemodynamic instability, active vomiting, bleeding, labor, severe pain, or acute need for hospital admission.
* Suicidal or homicidal ideation by chart review or on the Danger Assessment Scale for all assessed patients.
* No identifiable residence or contact phone number.
* Under arrest at the time of ED visit.
* Non-English speaking.
* Previously enrolled in the study.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2010-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Effectiveness of brief intervention for decreasing problem drinking and partner violence | Weekly for 3 months; then 6 and 12 months

SECONDARY OUTCOMES:
Assess impact of brief motivational intervention on IPV severity, alcohol quantity/frequency, self-rated health, health behaviors, quality of life, and relationship satisfaction | 3, 6, and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Karin V Rhodes, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Emergency Department, Hospital of the University of PA, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Rhodes KV, Rodgers M, Sommers M, Hanlon A, Crits-Christoph P. The Social Health Intervention Project (SHIP): protocol for a randomized controlled clinical trial assessing the effectiveness of a brief motivational intervention for problem drinking and intimate partner violence in an urban emergency department. BMC Emerg Med. 2014 Apr 18;14:10. doi: 10.1186/1471-227X-14-10. PMID 24742322
- [Derived] Hameed M, O'Doherty L, Gilchrist G, Tirado-Munoz J, Taft A, Chondros P, Feder G, Tan M, Hegarty K. Psychological therapies for women who experience intimate partner violence. Cochrane Database Syst Rev. 2020 Jul 1;7(7):CD013017. doi: 10.1002/14651858.CD013017.pub2. PMID 32608505
- [Derived] Rhodes KV, Rodgers M, Sommers M, Hanlon A, Chittams J, Doyle A, Datner E, Crits-Christoph P. Brief Motivational Intervention for Intimate Partner Violence and Heavy Drinking in the Emergency Department: A Randomized Clinical Trial. JAMA. 2015 Aug 4;314(5):466-477. doi: 10.1001/jama.2015.8369. PMID 26241598